CLINICAL TRIAL: NCT07158567
Title: Veterans' Intervention Blending NeuRomodulation and YogA for Chronic Low Back PaiN Treatment: VIBRANT
Brief Title: Veterans' Intervention Blending NeuRomodulation and YogA for Chronic Low BackPaiN Treatment: VIBRANT
Acronym: VIBRANT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RRD2-003-24W; I01 RD000449 (Other Grant/Funding Number: VA ORD RRDT POU AMP)
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain; Musculoskeletal Pain
Keywords: chronic low back pain; transcranial magnetic stimulation; TMS; neuromodulation; yoga; complementary and integrative health; musculoskeletal pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Transcranial Magnetic Stimulation; Yoga

STUDY DESIGN:
Intervention Model Description: single, blind, randomized, 3 parallel group design: (1) active-iTBS+yoga, (2) sham-iTBS+yoga, and (3) active-iTBS alone
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The PI, study statistician, intervention providers, and those collecting study data will be blind to treatment assignment. While participants may be able to discern whether or not they received iTBS alone because there is no yoga component (thus, the single blind), they may not be able to guess if they received active-iTBS+yoga vs. sham-iTBS. Participants will complete a blinding questionnaire after completion of the study intervention. After follow up, the study team will become unblinded to provide participants with the opportunity to complete their preferred intervention types. The study statistician will remained blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- active-iTBS+yoga (Experimental): real or active intermittent theta burst stimulation provided prior to participation in small group LoveYourBrain Yoga program class
  Interventions: Device: intermittent theta burst stimulation; Behavioral: LoveYourBrain Yoga Program
- sham-iTBS+yoga (Placebo Comparator): fake, inactive or sham intermittent theta burst stimulation (designed to look, sound and feel like real or active stimulation) provided prior to participation in small group LoveYourBrain Yoga program class
  Interventions: Device: intermittent theta burst stimulation; Behavioral: LoveYourBrain Yoga Program
- active-iTBS alone (Active Comparator): real or active intermittent theta burst stimulation alone (no yoga participation)
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive neuromodulatory treatment. TMS has been FDA cleared since 2008 for treatment resistant depression. It is now FDA cleared for a few other indications including migraine. Magnetic pulses are delivered through a coil placed on the scalp and when the magnetic field reaches brain cells, it changes to an electric current that can increase or decrease excitability depending on the treatment parameters. Intermittent theta burst stimulation (iTBS) is a type of patterned, excitatory TMS. iTBS only takes 3 minutes to deliver and is theorized to induce a window of neuroplasticity that lasts at least 1 hour. The Magventure with Magoption x100 Stimulator and associated coil the investigators are using can be set to deliver active (real) or sham (fake or inactive) TMS. The sham device is designed to look, sound and feel like real TMS.
  Other Names: transcranial magnetic stimulation (TMS), Magventure
Behavioral: LoveYourBrain Yoga Program — This yoga program is evidence-based, standardized and manualized. It is developed by the LoveYourBrain Foundation (www.loveyourbrain.com). Each yoga session includes 10 min of breathing exercises, 45 min of gentle yoga or stretching exercises, 15 min of guided meditation, and 20 min of facilitated discussion with psychoeducation, detailed in a manual to ensure standardization of program content across time and instructors.
  Other Names: yoga, hatha-based yoga
  Arms: active-iTBS+yoga; sham-iTBS+yoga

SUMMARY:
The objectives of this VA Merit application are to demonstrate efficacy of combined intermittent theta burst (iTBS) and yoga (iTBS+yoga) intervention on improving pain, function, analgesic use, self-efficacy, quality of life and well-being among Veterans with chronic low back pain (CLBP). This Merit project will directly benefit Veterans and VA Services by demonstrating efficacy of a new, non-medication treatment for Veterans with CLBP in need of non-opioid treatment options. Neuromodulation including iTBS is now offered at over 50 VA hospitals and yoga is among the complementary and integrative health programs being rolled out as a part of VAs Whole Health implementation efforts. Thus, should iTBS+yoga ultimately prove to be efficacious, VA facilities will be well-poised to offer this treatment. A novel, activity-based, non-medication treatment for Veterans with CLBP is of great need given the high prevalence of CLBP.

DETAILED DESCRIPTION:
Significance to VA: Chronic low back pain (CLBP) is the leading cause of disability worldwide and the most common location of chronic pain among Veterans. Medications are the treatment mainstay for CLBP and yet >50% of chronic pain patients receiving medications are treatment resistant. Lack of pain relief from medications can lead to non-prescription opioid use, opioid use disorder, and Veteran death from opioid overdose, which occurs at a higher rate than US Civilians. This Merit will directly benefit Veterans and VA Services by developing a new, neuromodulatory, non-opioid neurorehabilitation treatment for Veterans with CLBP who do not find existing options to be effective or preferable. Innovation and Impact: Yoga is an activity, and mindfulness-based behavioral intervention and is safe and recommended for CLBP. Given the room for improvement of available treatments and considering the life-threatening opioid epidemic, building an evidence base for novel, precise, non-medication approaches for pain management has high impact for VA Healthcare. The non-invasive treatment transcranial magnetic stimulation (TMS) applied to the motor cortex (M1) reduces pain and has remote effects including neuromodulation of pain pathways. Intermittent theta burst stimulation (iTBS), a type of patterned, excitatory TMS, increases M1 excitability. iTBS can prime the brain to boost the impact of interventions provided during this window of enhanced excitability. By activating the M1 through iTBS prior to participation in an evidence-based yoga program, the investigators theorize that iTBS will boost the effects of yoga resulting in improvements in pain, function and quality of life and these improvements will be sustained. The purpose of this Merit project is to demonstrate efficacy and additive effect of combined iTBS and yoga (iTBS+yoga) and vs. yoga or iTBS alone on improving pain, function, analgesic use, self-efficacy, quality of life (QOL) and well-being among Veterans with CLBP. This Merit is a natural progression of a VA RR&D-funded SPiRE suggesting that iTBS+yoga is safe, feasible, and acceptable among Veterans of all genders with CLBP and provides preliminary evidence of improvements from pre- to post-treatment in pain and QOL. The investigators will build on this evidence and add innovation by testing the additive effects of iTBS+yoga vs. yoga and iTBS each alone. For this Merit, the investigators will complete a randomized controlled trial among 3 groups of Veterans with CLBP receiving (1) active-iTBS+yoga, (2) sham-iTBS+yoga, or (3) active-iTBS alone. Specific Aims: Aim 1 will determine efficacy and sustainability of iTBS+yoga on pain, function, analgesic use, self-efficacy, QOL and well-being among Veterans with CLBP. Aim 2 will determine acceptability of iTBS+yoga for Veterans with CLBP. Exploratory Aim 3 will examine gender and common comorbidity measures as moderators of iTBS+yoga treatment effect. Methodology: The intervention will be provided in small group settings once a week for 6 weeks. Ac-tive- or sham-iTBS will be administered immediately prior to yoga. The investigators will be using an existing, evidence-based, manualized yoga program (LoveYourBrain Yoga). The investigators will collect outcome data related to pain, function, analgesic use, self-efficacy, QOL and well-being, as well as structural MRI data for iTBS neuronavigation. Path to Translation/Implementation: Completion of this Merit project will provide preliminary data for future applications focused on treatment responsiveness and a future larger scale multi-site pragmatic effectiveness study. This Merit project will directly benefit Veterans and VA Services by developing a new, non-pharmacological neurorehabilitation treatment for Veterans with CLBP in need of non-opioid treatment options. TMS is now offered at over 50 VA hospitals nationwide for treatment-resistant depression, and yoga is among the complementary and integrative health programs being rolled out as a part of VAs nation-wide Whole Health implementation efforts. Therefore, should iTBS+yoga ultimately prove to be efficacious and effective, VA facilities will be well-poised to offer this treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1 mo. stability in pain management strategies.
* 22+ years of age.
* Can read and speak English.
* Able to participate in strengthening, stretching, range of motion exercise via yoga as determined by study physician.
* Chronic Low Back Pain (CLBP): pain in the low back that persists for >6 months and is of moderate to severe intensity with a score of >5 on specific items on the BPI demonstrating disability of at least 20% on the Oswestry Disability Index (ODI).

Exclusion Criteria:

* Contraindications to iTBS/TMS (e.g. epilepsy, psychotic spectrum disorders [i.e. bipolar, schizophrenia], history of anoxic brain injury).
* Moderate to severe heart disease.
* Contraindications to MRI (e.g., claustrophobia, implanted ferromagnetic device such as pacemaker or cardiac defibrillator).
* Pain believed to be associated with cardiac or ischemic conditions.
* Epilepsy, active seizure disorder, personal history of a seizure or individuals with a family history of epilepsy or seizure in a first degree relative.
* Current prescription of psychostimulants (e.g., amphetamines), anticholinergics, tricyclic antidepressants, and antipsychotics or other medications that may increase their risk of having seizures.
* Intracranial lesion.
* History of ischemic or hemorrhagic stroke.
* History of moderate to severe TBI.
* History of or current psychosis not due to an external cause (e.g., due to illicit drug use).
* Other neurological conditions (e.g., neurodegenerative disorders).
* Active suicidal ideation with Columbia Suicide Severity Rating Scale(CSSRS) 3 .
* Are pregnant or nursing.
* Within 12 weeks of a major surgery/operation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Pain Severity | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The Brief Pain Inventory is a self-report measure of pain symptoms throughout the body. It has 4 main items related to pain severity and each item is scored on a scale of 0 to 10 with 0 meaning no pain (better), and 10 meaning pain as bad as you can imagine (worse). Minimum (best) score would be 0 and maximum (worst) score would be 40.
Brief Pain Inventory - Pain Interference | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The Brief Pain Inventory is a self-report measure of pain symptoms throughout the body. t has 7 main items related to pain interference and each item is scored on a scale of 0 to 10 with 0 meaning "Does not interfere", and 10 meaning "Completely Interferences". Minimum (best) score would be 0 and maximum (worst) score would be 70.

SECONDARY OUTCOMES:
PROMIS Pain Interference - Short Form 6b | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The Pain Interference - Short Form 6b is a 6-item self-report measure of pain interference. Each item is scored on a scale of 1 "not at all" (better) to 5 "very much" (worse). Minimum (best) possible raw score would be 6 and maximum (worst) possible raw score would be 30. Raw scores are converted with a conversion chart from the manual to a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10.
PROMIS Physical Function with Mobility Aid | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The Physical Function with Mobility Aid is an 11-item self-report measure of daily life functioning and mobility. Each item is scored on a scale of 5 "without any difficulty" (best) to 1 "unable to do" (worst). The maximum (best) possible raw score is 55 and the minimum (worst) possible raw score is 11. Raw scores are converted with a conversion chart from the manual to a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10.
Wellbeing Signs Tool | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The well being signs tool is a self-report measure that starts with an open ended question of "what matters most to you in your life right now?" followed by 3 items on a scale of 0 to 10 with 0 being the worst and 10 being the best wellbeing. The minimum (worst) possible score is 0 with the maximum (best) possible score of 30.
Pain Self-Efficacy Questionnaire | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The Pain Self-Efficacy Questionnaire is a self-report measure that asks about confidence in doing things at the present time despite the pain. It has 2 items and each item is has a scale of 0 to 6 with 0 being "not at all confident" (worst) and 6 being "completely confident" (best). The total minimum (worst) possible raw score would be 0 and total maximum (best) possible raw score would be 12. A person with a score of 5 or less might be considered in need of help with their confidence in functioning in the presence of their pain. A score of 8 or higher reflects a desirable level of pain self-efficacy or confidence in functioning in the presence of pain.
Veterans Rand 36 Item Health Survey (VR-36) | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The VR-36 is a 36-item self-report measure of health-related quality of life. The VR-36 yields mental and physical component scores (MCS and PCS), with higher scores indicating better health-related quality of life.
Pain Catastrophizing Scale (PCS) | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  The pain catastrophizing scale is a 13-item self report measure that asks about the types of thoughts and feelings associated with pain. The participant indicates the degree to which they think they have these thoughts and feelings when they are in pain on a scale of 0 "not at all" (best) to 4 "all the time" (worst). The minimal (best) possible score is a 0 and the maximum (worst) possible score is a 52. Item scores are summed into a total score (PCS-T) and 3 subscale scores rumination (PCS-R, Items 8,9,10 and 11), magnification (PCS-M, Items 6,7,13), and helplessness (PCS-H, Items 1,2,3,4,5, and 12). A total score above 30 indicates clinically relevant level of catastrophizing.
analgesic use | Baseline (Pre-intervention, Endpoint (after last iTBS+yoga treatment, approximately 6 weeks), Follow-Up at 1 week, 2 weeks, 6 weeks and 6 months post-treatment
  A medication inventory will be completed including opioids, other prescription and over the counter pain medications. The medication, dose, frequency and mode (e.g., oral, intramuscular injection, etc..) will be recorded. We will use total dosage over the 6 week study intervention and 6 month follow up period of medications as the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Herrold, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The NICHD Data and Specimen Hub (DASH) is a centralized resource that allows researchers to share and access de-identified data — https://dash.nichd.nih.gov